CLINICAL TRIAL: NCT03947658
Title: Influence of Prosthetic Restorative Treatment Timing on Gingival Margin of Teeth After Surgical Crown Lengthening: a Randomized Controlled Pilot Study.
Brief Title: Influence of Restorative Timing on Crown Lengthening Outcome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Tsachouridou Ioanna, DDS, MSc in Periodontology and Implant Biology, Private practice, Thessaloniki, Greece, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30/03-05-2017
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Crown Lengthening
Keywords: surgical; prosthetic restoration; gingiva; surgical flaps; stents

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Six weeks group (Experimental): Prosthetic restoration started 6 weeks after surgical crown lengthening
  Interventions: Procedure: Surgical crown lengthening
- Fourteen weeks group (Experimental): Prosthetic restoration started 14 weeks after surgical crown lengthening
  Interventions: Procedure: Surgical crown lengthening

INTERVENTIONS:
Procedure: Surgical crown lengthening — Surgical lengthening of teeth with short clinical crown and prosthetic rehabilitation

SUMMARY:
Setting the restorative margins for teeth with short clinical crowns is challenging and crown lengthening surgery (CLS) is often necessary. The aim of this study was to assess the influence of prosthetic restorative treatment timing on gingival margin location of teeth after crown lengthening surgery.

Eighteen patients requiring CLS were enrolled in the study and divided into two groups depending on the timing of prosthetic rehabilitation, at 6 or fourteen weeks after CLS.Clinical parameters were recorded around treated and neighboring teeth with adjacent and non-adjacent sites at 6 and 14 weeks after surgery as well as three and six months after prosthesis delivery. Alveolar ridge changes were assessed via digital X-rays.Soft tissue healing and the final treatment outcome were assessed by both patients and prosthodontists.

DETAILED DESCRIPTION:
Twenty patients selected from those referred to the Department of Periodontics for crown lengthening surgery were enrolled in the study (9 females, 11 males, 19-65 years old, mean age:45.2) Patients were randomly assigned to one of the two experimental groups. For the first group of patients (A), prosthetic restoration started 6 weeks whereas for the second group (B)14 weeks after surgery. After recording of pre-surgical measurements, intrasulcular or internal bevel incisions were performed buccally and lingually, and full-thickness mucoperiosteal flaps were raised. Buccal flaps were reflected to a level beyond the mucogingival junction. The osseous crest and subgingival tooth structure were exposed. The osseous resection was performed after considering the amount of additional tooth structure required for restorative purpose and the preoperative Supracrestal Tissue Attachment at each site with hand and rotary instruments in a manner of establishing positive bone architecture. After root planing, suturing of the surgical sites was performed. The flap margins were placed at or apical to the anticipated crown margin after suturing and as far from the osseous crest as possible and necessary postoperative instructions were given. Patients were recalled 1 week post-surgery for suture removal, oral hygiene reinforcement and healing assessment. Healing was also evaluated at the end of the second post-operative week. All patients were reevaluated at 3 and 6 months after the prosthesis delivery.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years,
* periodontally healthy or periodontally treated subjects with Plaque scores ≤15% & GI ≤15%
* each patient could participate with one tooth only,
* non-smokers or smokers of less than 5 cigarettes per day,
* target tooth should be surrounded by both the adjacent teeth which should not be restored,
* provisional and final prosthetic margins should not extend subgingivally,
* in case of fracture this should be radiographically detectable,
* if a root canal treatment was necessary it should have been completed at least 6 months earlier.
* both anterior and posterior teeth included.

Exclusion Criteria:

* the presence of syndromes affecting bone metabolism,
* any kind of contraindication for periodontal surgery,
* pregnancy or lactation,
* no compliance with re-examinations or oral hygiene performance
* cases where gingivectomy or apically repositioned flap without osseous resection were indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Relative gingival margin location change | 6 months after prosthesis delivery (30 to 38 weeks after surgery)
  The relative position of free gingival margin as measured from an individualized reference stent in millimeters

SECONDARY OUTCOMES:
Pocket depth | before surgery, immediately after surgery, 6 weeks after surgery, 14 weeks after surgery,at prosthesis delivery, 3 and 6 months after prosthesis delivery
  Distance from gingival margin-the base of the pocket in millimeters
Relative clinical attachment loss | before surgery, immediately after surgery, 6 weeks after surgery, 14 weeks after surgery, at prosthesis delivery, 3 and 6 months after prosthesis delivery
  Distance from reference stent to the base of the pocket in millimeters
Plaque index | before surgery, immediately after surgery, 6 weeks after surgery, 14 weeks after surgery, at prosthesis delivery, 3 and 6 months after prosthesis delivery
  The number of sites presenting with dental plaque appositions
Gingival bleeding index | before surgery, immediately after surgery, 6 weeks after surgery, 14 weeks after surgery, at prosthesis delivery, 3 and 6 months after prosthesis delivery
  The number of sites presenting with bleeding on probing

OTHER OUTCOMES:
Reference stent to the osseous crest before surgery | Before surgery
  The distance between the reference stent to the osseous crest in millimeters
Reference stent to the osseous crest after surgery | Immediately after surgery completion
  The distance from the reference stent to the osseous crest in millimeters
Gingival margin after suturing. | Immediately after surgery completion
  The distance between the reference stent and the free gingival margin in millimeters
Radiographic change of alveolar crest | 6 months after prosthesis delivery (30 to 38 weeks after surgery)
  The root apex was used as a reference point and linear measurements from the reference point to the osseous crest of the target-tooth and the adjacent teeth mesially and distally on digital x-rays in millimeters
Early wound healing index | At the end of the first and second week after surgery
  A four-grade soft tissue healing evaluation with the use of Early Healing Index by Wachtel et al 2003. 1 indicates complete flap closure without fibrin line in the interproximal area; 2: complete flap closure with fine fibrin line in the interproximal area;3: complete flap closure with fibrin clot in the interproximal area; 4: incomplete flap closure with partial necrosis of the interproximal tissue 5: incomplete flap closure - complete necrosis of the interproximal tissue
Patient pain and discomfort | End of first week after surgery
  Questionnaire of 6 questions asking about pain, discomfort and swelling experienced by the patient due to surgery. The participant responds by choosing an answer from a scale is graded from 1 to 10 with 1 representing the worst and 10 the best answer.
Patient satisfaction from prosthetic restoration | after the end of prosthetic restoration (8 to 16 weeks after surgery)
  Questionnaire of 3 questions for the evaluation of patients' satisfaction from the aesthetics and function of the restoration. The participant responds by choosing an answer from a scale is graded from 1 to 10 with 1 representing the worst and 10 the best answer.
Prosthodontist's satisfaction | after the end of prosthetic restoration (8 to 16 weeks after surgery)
  Questionnaire of 4 questions for the evaluation of prosthodontists' satisfaction from the outcome of the surgical intervention in terms of availability of tooth structure, tooth mobility, bone support adequacy and soft tissue aesthetics.The prosthodontist responds by choosing an answer from a scale is graded from 1 to 10 with 1 representing the worst and 10 the best answer.

REFERENCES:
- [Derived] Malamoudi GA, Tsachouridou I, Menexes G, Mikrogeorgis G, Tortopidis D, Tsalikis L. Pre-restorative crown lengthening surgery: influence of restorative treatment timing on clinical outcomes-a pilot study. Oral Maxillofac Surg. 2024 Mar;28(1):253-267. doi: 10.1007/s10006-023-01138-6. Epub 2023 Jan 25. PMID 36695965